CLINICAL TRIAL: NCT02268617
Title: Immediate Effects of Treadmill Walking in Individuals With Dementia With Lewy Bodies and Huntington's Disease
Brief Title: Treadmill Walking in Individuals With Dementia With Lewy Bodies and Huntington's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Anne Kloos, Associate Clinical Professor, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012H0385
Record Dates: First submitted 2014-10-10; First posted 2014-10-20 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Huntington Disease; Lewy Body Disease
Keywords: Treadmill; Walking; Gait; Exercise
MeSH Terms: conditions — Huntington Disease; Lewy Body Disease; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treadmill Walking (Experimental): All subjects will walk on treadmill for a total of 20 minutes.
  Interventions: Other: Treadmill Walking

INTERVENTIONS:
Other: Treadmill Walking — Following instructions and familiarization with the treadmill, participants will walk on the treadmill for 20 minutes total with rest periods as needed. Treadmill speed will be set at each participant's overground comfortable walking speed for the first 5 minutes, provided that they can walk safely. If necessary the speed will be lowered until a safe gait is achieved. After 5 minutes the speed will be incrementally increased by10% each 5 minutes (3 times) as long as a safe gait (i.e., no abnormal vital signs, excessive effort, or loss of balance occurrences) can be maintained. If the gait pattern becomes unsafe or more abnormal the speed will revert to the previous safe speed and be maintained at this level until the end of training session.

SUMMARY:
Individuals with Dementia with Lewy Bodies (DLB) and Huntington's disease (HD) experience balance and walking problems that lead to falls. Treadmill walking has demonstrated improvements in balance and walking and fall risk in individuals with Parkinson's disease (PD), suggesting that it may be beneficial for individuals with DLB and HD. In PD subjects, changes in gait parameters have been noted after only one treadmill training session. The investigators propose a pilot study to investigate the safety, feasibility, and utility to improve mobility and fall risk of a single session of treadmill walking in individuals with DLB and HD.

DETAILED DESCRIPTION:
Several studies using HD animal models have shown that HD mice housed in enriched environments or in cages with running wheels that stimulated physical activity demonstrated a delayed onset and/or slowed decline in motor function compared to mice in non-enriched environments (van Dellen et al. 2000, 2008; Spires et al., 2004). Evidence suggests that aerobic exercise may have neuroprotective effects and helps the elderly and individuals with neurodegenerative diseases to maintain better cognitive and motor function than those who are inactive. More specifically, there is strong evidence from animal and human trials in neurological populations (i.e., Parkinson's Disease, spinal cord injury, and stroke) that treadmill training can improve walking and motor function. Immediate effects of a single-session of treadmill walking in the Parkinson's Disease population were improved over-ground gait measures (i.e., gait speed, stride length, double support percent, stride variability) and longer term treadmill training studies demonstrated additional improvements in Unified Parkinson Disease Rating Scale scores, fall risk, and health-related quality of life (Herman et al., 2008). This study builds upon foundational knowledge gained in animals and other neurologic populations to determine the feasibility, safety and possible immediate benefit of treadmill walking in individuals with HD.

The primary purpose of this pilot study is to investigate the the safety, feasibility and utility of a single 20-minute session of treadmill walking to improve gait parameters in ambulatory individuals with DLB and HD. Secondarily we will explore the effects of treadmill walking on mobility, fall risk, and motor coordination. Based on previous studies utilizing a single-session of treadmill training in the PD population, we hypothesize that treadmill walking will improve overground spatiotemporal gait parameters (gait speed, stride length, double support percent, and stride-to-stride variations in gait) in individuals with DLB and HD (Pohl et al., 2003; Frenkel-Toledo et al., 2005; Bello et al., 2008).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Huntington's disease or Dementia with Lewy Bodies,
* the ability to ambulate 80 feet without assistance, and
* the ability to provide informed consent and understand directions.

Exclusion Criteria:

* presence of any clinically significant musculoskeletal or neurological disease that would affect gait.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-02; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Vital signs | Within 24 hours
  Blood pressure, heart rate, and rating of perceived exertion will be measured before, during, and after treadmill walking.

SECONDARY OUTCOMES:
Spatiotemporal gait measures | within 24 hours
  Spatiotemporal gait parameters will be measured using a computerized system, a 4.88 meter electronic carpet equipped with sensors that record footfalls and communicate the information to a computer software program.
Timed Up and Go Test | Within 24 hours
  Mobility and fall risk will be measured using the Timed Up and Go Test (TUG) that includes standing up from a chair, walking 3 meters, turning and returning to sitting in the chair.
Q-motor testing | Within 24 hours
  Motor coordination will be measured using force-transducer based measurement of grip forces during grasping and holding an object and of tapping forces and tap interval variability during fast repetitive finger and foot tapping.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Kloos, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Physical Therapy Division, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bello O, Sanchez JA, Fernandez-del-Olmo M. Treadmill walking in Parkinson's disease patients: adaptation and generalization effect. Mov Disord. 2008 Jul 15;23(9):1243-9. doi: 10.1002/mds.22069. PMID 18464281
- [Background] Bechtel N, Scahill RI, Rosas HD, Acharya T, van den Bogaard SJ, Jauffret C, Say MJ, Sturrock A, Johnson H, Onorato CE, Salat DH, Durr A, Leavitt BR, Roos RA, Landwehrmeyer GB, Langbehn DR, Stout JC, Tabrizi SJ, Reilmann R. Tapping linked to function and structure in premanifest and symptomatic Huntington disease. Neurology. 2010 Dec 14;75(24):2150-60. doi: 10.1212/WNL.0b013e3182020123. Epub 2010 Nov 10. PMID 21068430
- [Background] Bilney B, Morris ME, Churchyard A, Chiu E, Georgiou-Karistianis N. Evidence for a disorder of locomotor timing in Huntington's disease. Mov Disord. 2005 Jan;20(1):51-7. doi: 10.1002/mds.20294. PMID 15390128
- [Background] Churchyard AJ, Morris ME, Georgiou N, Chiu E, Cooper R, Iansek R. Gait dysfunction in Huntington's disease: parkinsonism and a disorder of timing. Implications for movement rehabilitation. Adv Neurol. 2001;87:375-85. No abstract available. PMID 11347241
- [Background] Frenkel-Toledo S, Giladi N, Peretz C, Herman T, Gruendlinger L, Hausdorff JM. Treadmill walking as an external pacemaker to improve gait rhythm and stability in Parkinson's disease. Mov Disord. 2005 Sep;20(9):1109-14. doi: 10.1002/mds.20507. PMID 15929090